CLINICAL TRIAL: NCT03409328
Title: Understanding and Reducing HIV Risk Behavior and Substance Use Among Self-identified Bisexual Adolescent Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rosalind Franklin University of Medicine and Science (Other)
Responsible Party: Principal Investigator, Brian A. Feinstein, Associate Professor, Rosalind Franklin University of Medicine and Science
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 9481383
Record Dates: First submitted 2018-01-11; First posted 2018-01-24 (Actual); Results first posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: HIV/AIDS; Substance Use; Bisexuality
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Substance-Related Disorders; Bisexuality | interventions — Seroconversion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIV and substance use prevention (Experimental): Participants in the intervention condition will receive an HIV and substance use prevention program for self-identified bisexual adolescent men. The intervention content will be developed through formative research during the initial phase of the study.
  Interventions: Behavioral: HIV and substance use prevention
- Waitlist (No Intervention): The control condition will be a waitlist.

INTERVENTIONS:
Behavioral: HIV and substance use prevention — The intervention content will be developed through formative research during the initial phase of the study. However, the intervention will address: bisexual-inclusive sexual health education, unique influences of risk behavior among bisexual adolescents, and skills to cope with bisexual stigma and to increase acceptance of one's bisexual identity.
  Arms: HIV and substance use prevention

SUMMARY:
Young gay, bisexual, and other men who have sex with men (MSM) are disproportionately affected by HIV. Despite this burden, most HIV prevention interventions target adult MSM (most of whom identify as gay) and heterosexual youth, creating an urgent need for interventions for gay and bisexual adolescents. Further, self-identified bisexual men, especially adolescents, have been neglected in research. Therefore, little is known about factors that drive engagement in risk behavior among self-identified bisexual adolescent men. The goals of this study are to: (1) examine factors that drive engagement in HIV risk behavior and substance use among self-identified bisexual adolescent men; and (2) develop and pilot test a tailored HIV and substance use prevention intervention for this population.

DETAILED DESCRIPTION:
Young gay, bisexual, and other men who have sex with men (MSM) are disproportionately affected by HIV. Despite this burden, most HIV prevention interventions target adult MSM (most of whom identify as gay) and heterosexual youth, creating an urgent need for interventions for gay and bisexual adolescents. Further, self-identified bisexual men, especially adolescents, have been neglected in research. This is a critical problem because: (1) there are as many, if not more, bisexual adolescent men than gay adolescent men; (2) bisexual adolescent men engage in several HIV risk behaviors more than their gay peers; (3) bisexual adolescent men are at increased risk for substance use-a robust risk factor for HIV; and (4) bisexual men face unique HIV prevention issues. Given that bisexual men are rarely included in research and most existing research on them focuses on "behaviorally bisexual" adult men, little is known about factors that drive engagement in risk behavior among self-identified bisexual adolescent men. Attending to bisexual identity is critical to reducing HIV and substance use, because bisexuality is highly stigmatized and stigma-related stressors (e.g., concerns about disclosing one's bisexual identity) impact sexual behavior, substance use, and healthcare utilization. Interventions are also more effective when tailored to populations, underscoring the need for an intervention for self-identified bisexual adolescent men. The goals of this study are to: (1) examine factors that drive engagement in HIV risk behavior and substance use among self-identified bisexual adolescent men; and (2) develop and pilot test a tailored HIV and substance use prevention intervention for this population. In Phase 1, interviews will be conducted with 60 diverse self-identified bisexual adolescent men ages 14-17 focused on sexual identity, sexual decision-making, substance use motivations, and intervention preferences/barriers. In Phase 2, a tailored intervention will be developed using findings from Phase 1. In Phase 3, feasibility, acceptability, and preliminary efficacy will be tested in a pilot randomized trial (N = 60) with a waitlist control and one-month follow-up. In sum, self-identified bisexual adolescent men are at increased risk for HIV and substance use, but little is known about factors that drive their engagement in risk behavior. By focusing on self-identified bisexual adolescent men-an underrepresented, health disparity population-this study can identify prevention targets and reduce disparities in HIV and substance use.

ELIGIBILITY:
Inclusion Criteria:

* Age 14-17
* Identifies as male
* Identifies as bisexual or another non-monosexual identity (e.g., pansexual)
* HIV-negative (self-report)
* Fluent in English
* Lives in United States

Exclusion Criteria:

* Does not meet inclusion criteria

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Participants must self-identify as male regardless of their sex assigned at birth.
Enrollment: 60 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian A Feinstein, PhD, Principal Investigator — Rosalind Franklin University of Medicine and Science
Locations (1):
- Rosalind Franklin University of Medicine and Science, North Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Investigators can contact the PI to discuss potential use of the data for purposes other than those specified in the specific aims. These requests will be considered by the PI on a case-by-case basis to ensure that all investigators are qualified and that the data will be used in a responsible and ethical manner. If the data are shared, a data sharing agreement will be developed and all shared data will be de-identified.

RESULTS

PARTICIPANT FLOW:
Groups:
- B*SMART: B*SMART is an online HIV and substance use prevention intervention for self-identified bisexual adolescent men. It includes 90 minutes of content, which can be completed in a single session or across multiple sessions. Participants had one month to complete the intervention. It includes 4 modules that participants can navigate in their preferred order. Within each module, information is presented via text, audio, video, and activities. The modules cover topics related to (1) sexual orientation and gender identity (e.g., coming out, reducing internalized stigma, positive aspects of being bisexual), (2) sexual activity, pleasure, and consent, (3) HIV/STI (e.g., types, level of risk associated with different sexual activities, types of protection, the influence of substance use), and (4) healthy relationships (e.g., different relationship configurations, effective communication).
- Waitlist: The control condition was a waitlist.
Period: Overall Study
Arm/Group | B*SMART | Waitlist
Started | 31 | 29
Completed | 25 | 26
Not Completed | 6 | 3
Not completed — Lost to Follow-up | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | B*SMART | Waitlist | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.94 (1.03) | 15.93 (.96) | 15.93 (.99)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex/gender: Cisgender boys | 23 | 22 | 45
  Sex/gender: Transgender boys | 8 | 7 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: White (non-Hispanic) | 17 | 16 | 33
  Race/ethnicity: Black (non-Hispanic) | 1 | 1 | 2
  Race/ethnicity: Hispanic | 8 | 7 | 15
  Race/ethnicity: Other (non-Hispanic) | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 31 | 29 | 60
HIV status [Count of Participants; unit: Participants]
  Negative | 4 | 5 | 9
  Unknown | 27 | 24 | 51

OUTCOME MEASURES:

1. Primary Outcome: Retention
Description: Retention from enrollment through the 1-month follow-up assessment.
Time Frame: Up to 2 months (participants in the intervention condition had 1-month to complete the intervention and the follow-up assessment was 1-month later; participants in the control condition waited for 1-month and then completed the follow-up assessment).
Measure: Count of Participants; unit: Participants
Arm/Group | B*SMART | Waitlist
Number analyzed (Participants) | 31 | 29
Participants | 25 | 26

2. Primary Outcome: Acceptability
Description: Acceptability was measured with an adapted version of the Abbreviated Acceptability Rating Profile. Scores ranged from 0-4. Higher scores represent greater acceptability.
Time Frame: Post-intervention
Population: Of the 31 participants in the intervention condition, 24 completed the intervention and 16 completed the post-intervention acceptability survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | B*SMART
Number analyzed (Participants) | 16
score on a scale | 3.62 (.36)

3. Secondary Outcome: HIV Knowledge
Description: Participants were asked 12 true/false questions to assess their HIV knowledge. Values ranged from 0-12. Higher scores represent greater HIV knowledge.
Time Frame: 1-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | B*SMART | Waitlist
Number analyzed (Participants) | 25 | 26
score on a scale | 9.32 (1.07) | 6.85 (1.91)
Statistical Analysis 1: Comparison: B*SMART vs Waitlist; Test type: Other; p < .001, ANCOVA; The ANCOVA controlled for baseline levels of the outcome; F = 38.44

4. Secondary Outcome: Sexually Transmitted Infection (STI) Knowledge
Description: Participants were asked 12 true/false questions to assess their STI knowledge. Scores ranged from 0-12. Higher scores represent greater STI knowledge.
Time Frame: 1-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | B*SMART | Waitlist
Number analyzed (Participants) | 25 | 26
score on a scale | 7.75 (2.59) | 5.70 (2.48)
Statistical Analysis 1: Comparison: B*SMART vs Waitlist; Test type: Other; p = .013, ANCOVA; The ANCOVA controlled for baseline levels of the outcome; F = 6.69

5. Secondary Outcome: Condom Use Intentions
Description: Participants were asked eight questions to assess their intentions to use condoms. Scores ranged from 1-4. Higher scores represent greater condom use intentions.
Time Frame: 1-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | B*SMART | Waitlist
Number analyzed (Participants) | 25 | 26
score on a scale | 3.62 (.51) | 3.33 (.56)
Statistical Analysis 1: Comparison: B*SMART vs Waitlist; Test type: Other; p = .029, ANCOVA; The ANCOVA controlled for baseline levels of the outcome; F = 5.07

6. Secondary Outcome: Condom Use Self-efficacy
Description: Participants were asked eight or nine questions to assess their condom use self-efficacy (cisgender participants received one question that transgender participants did not receive). Scores ranged from 1-7. Higher scores represent greater condom use self-efficacy.
Time Frame: 1-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | B*SMART | Waitlist
Number analyzed (Participants) | 25 | 26
score on a scale | 6.08 (1.08) | 5.89 (.91)
Statistical Analysis 1: Comparison: B*SMART vs Waitlist; Test type: Other; p = .542, ANCOVA; The ANCOVA controlled for baseline levels of the outcome; F = 0.38

7. Secondary Outcome: Internalized Stigma and Identity Affirmation
Description: Internalized stigma and identity affirmation were measured with the Bisexual Identity Inventory. Scores ranged from 1-7. Higher scores represent greater internalized stigma or identity affirmation.
Time Frame: 1-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | B*SMART | Waitlist
Number analyzed (Participants) | 25 | 26
score on a scale
  Internalized stigma | 2.56 (1.53) | 2.86 (1.32)
  Identity affirmation | 5.47 (1.54) | 5.50 (.96)
Statistical Analysis 1: Comparison: B*SMART vs Waitlist; The outcome for this analysis is internalized stigma; Test type: Other; p = .084, ANCOVA; The ANCOVA controlled for baseline levels of the outcome; F = 3.12
Statistical Analysis 2: Comparison: B*SMART vs Waitlist; The outcome for this analysis is identity affirmation; Test type: Other; p = .417, ANCOVA; The ANCOVA controlled for baseline levels of the outcome; F = 0.67

8. Secondary Outcome: Condomless Sex
Description: Participants were asked a series of questions about their sexual activity and condom use from the HIV-Risk Assessment for Sexual Partnerships. Condomless sex (anal or vaginal) was treated as a dichotomous variable (0 = none, 1 = any).
Time Frame: 1-month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | B*SMART | Waitlist
Number analyzed (Participants) | 25 | 26
Participants
  Engaged in condomless sex | 2 | 2
  Did not engage in condomless sex | 23 | 24

9. Secondary Outcome: Substance Use
Description: Participants were asked a series of questions about their alcohol and drug use. Outcomes included binge drinking and marijuana use. Outcomes were dichotomous (any vs. none).
Time Frame: 1-month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | B*SMART | Waitlist
Number analyzed (Participants) | 25 | 26
Participants
  Binge drinking | 1 | 1
  Marijuana use | 6 | 6

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for up to 2 months.
Arm/Group | B*SMART | Waitlist
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/29
Other Adverse Events (participants affected / at risk) | 0/31 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT03409328/Prot_SAP_000.pdf